CLINICAL TRIAL: NCT01968265
Title: A Randomized, Double Blind, Placebo-Controlled, Phase 2 Study to Assess the Safety, Tolerability and Efficacy of ISIS 426115 (an Antisense Glucocorticoid Receptor Antagonist) Administered Subcutaneously Once Weekly for 6 Weeks to Patients With Type 2 Diabetes Mellitus Being Treated With Metformin
Brief Title: Safety, Tolerability and Efficacy of ISIS-GCCRRx in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS 426115-CS2; 2013-002172-40 (EudraCT Number)
Record Dates: First submitted 2013-10-18; First posted 2013-10-24 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- ISIS-GCCRRx (Active Comparator)
  Interventions: Drug: ISIS-GCCRRx

INTERVENTIONS:
Drug: ISIS-GCCRRx — 3 doses on alternate days during the first week and then once weekly for 5 weeks + daily metformin
  Arms: ISIS-GCCRRx
Drug: Placebo — 3 doses on alternate days during the first week and then once weekly for 5 weeks + daily metformin
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of ISIS-GCCRRx in combination with metformin versus placebo + metformin

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 to 75
* BMI greater than or equal to 25
* HbA1c greater than or equal to 7.5% and less than or equal to 10.5%
* Type 2 Diabetes Mellitus and on stable dose of oral metformin
* Agree to conduct home-based (fasted) blood glucose testing as directed

Exclusion Criteria:

* Clinically significant abnormalities in medical history or physical exam
* Show evidence of uncorrected hypothyroidism or hyperthyroidism hormone results
* History of renal transplantation or renal dialysis
* History of liver disease
* History of greater than 3 episodes of severe hypoglycemia within 6 months of screening
* Use of oral anti-diabetic medication other than metformin within 3 months of screening
* Use of medications that may affect plasma glucose levels (including systemic glucocorticoids), systemic steroids, corticosteroids, antiglucocorticoid therapies including mifepristone and ketoconazole (topical cream and systemic), immunosuppressive medications, somatostatin analogues or ACTH therapy within 3 months of screening
* History of diabetic ketoacidosis
* Current or previous diagnosis of Gilbert's disease
* Any other significant illness or condition that may interfere with the patient participating or completing the study
* Inability or unwillingness to comply with protocol or study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The effect of ISIS-GCCRRx on serum fructosamine | 7 Weeks
  Change from Baseline to Week 7

SECONDARY OUTCOMES:
The safety of ISIS-GCCRRx | 18 Weeks
  By determining the incidence, severity, adverse effects, and changes in laboratory evaluations
The tolerability of ISIS-GCCRRx | 18 Weeks
  By determining the incidence, severity, adverse effects, and changes in laboratory evaluations

CONTACTS AND LOCATIONS:
Locations (13):
- Canada (6):
  - Isis Investigative Site, Red Deer, Alberta
  - Isis Investigative Site, Penticton, British Columbia
  - Isis Investigative Site, Cornwall, Ontario
  - Isis Investigative Site, Courtice, Ontario
  - Isis Investigative Site, Greater Sudbury, Ontario
  - Isis Investigative Site, Montreal, Quebec
- Romania (3):
  - Isis Investigative Site, Bucharest, Bucharest
  - Isis Investigative site, Bucharest, Bucharest
  - Isis Investigative Site, Cluj-Napoca, Cluj
- South Africa (4):
  - Isis Investigative Site, Bloemfontein, Free State
  - Isis Investigative Site, Benoni, Gauteng
  - Isis Investigative Site, Soweto, Gauteng
  - Isis Investigative Site, Somerset West, Western Cape